CLINICAL TRIAL: NCT05492435
Title: Changes in EEG Microestates After Combined Treatment od Tdcs and Dual-task Training in Stroke Patients: a Cross-roads, Sham-controlled,Double-blind Clinical Trial
Brief Title: CEEG Changes After Tdcs and Dual-task Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Andrade, Dra, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: microstates_stroke
Record Dates: First submitted 2022-07-19; First posted 2022-08-08 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Electroencephalogram
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- m1 stimulation + dual task training (Experimental): participants will receive real current over the primary motor area (M1)
  Interventions: Device: transcranial direct current stimulation
- stimulation in M1 and DLPF + dual task training (Experimental): participants will receive real current over the M1 and over the dorsolateral prefrontal area (DLPFC)
  Interventions: Device: transcranial direct current stimulation
- sham stimulation + dual task training (Sham Comparator): Participants will receive simulated stimulation
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS can regulate cortical excitability by influencing membrane polarity, where anodic current increases excitability and cathodic current reduces excitability. Therefore, in post-stroke patients when the anode is applied to the cerebral hemisphere ipsilesional to the lesion or the cathode to the contralesional hemisphere, the balance between the interhemispheres tends to be restored.

SUMMARY:
Stroke has been considered one of the main causes of long-term disability in the adult population. Technological advances in the neurological area have been observed in the last decades, which accentuates the interest in promoting non-invasive stimulation techniques, capable of modulating brain polarity, where among these techniques is the transcranial direct current stimulation - tDCS. Previous studies analyzed by systematic reviews suggest that the effects of tDCS may vary between individuals, where some stroke patients may not receive any additional benefit from the therapy. Thus, it is necessary to use a biomarker that can choose those that will possibly benefit from the electric current. Therefore, the aim of this study is to identify the dynamics of EEG microstates after tDCS and dual-task training in subjects after chronic stroke, as well as to assess how microstate parameters in stroke patients are altered by tDCS and dual-task training. at three different moments (Stimulation in M1 + dual-task training; Stimulation in M1 and DLPF + dual-task training; Sham stimulation) and to observe whether the microstates encode information that reflects the motor and/or cognitive capacity of these patients.

DETAILED DESCRIPTION:
Cerebrovascular Accident (CVA) has been considered one of the main causes of long-term disability in the adult population. Stroke usually causes deficits such as asymmetrical muscle weakness between limbs, impaired proprioceptive ability, sensory loss, vision problems, and spasticity. In post-stroke patients, it is believed that the interhemispheric balance may be altered as a result of brain injury, the theory of interhemispheric competition is widely used as a theoretical basis for the application of non-invasive neuromodulatory techniques. Technological advances in the neurological field have been seen in recent decades, which accentuates the interest in promoting non-invasive stimulation techniques, capable of modulating brain polarity, where among these techniques is transcranial direct current stimulation - tDCS. Previous studies analyzed by systematic reviews suggest that the effects of tDCS may vary between subjects, where some stroke patients may not receive any additional benefit from the therapy. Thus, it is necessary to use a biomarker that can choose those who will possibly benefit from the electric current. Therefore, the aim of this study is to identify the dynamics of EEG microstates after tDCS and dual-task training in subjects after chronic stroke, as well as to assess how microstate parameters in stroke patients are altered by tDCS and dual-task training at three different times (Stimulation in M1 + dual-task training; Stimulation in M1 and DLPF + dual-task training; Sham stimulation) and observe whether the microstates encode information that reflects the motor and/or cognitive capacity of these patients. For this, a clinical trial, sham-controlled, double-blind and randomized, of crossover type, involving patients with stroke in chronic stage will be carried out. Participants will be submitted to three sessions, each session consisting of a different condition, namely: first condition (anodic tDCS) participants will receive real current over the primary motor area (M1); second condition (dualsite tDCS) participants will receive real current over M1 and dorsolateral prefrontal area (DLPFC) and third condition (sham tDCS) participants will receive simulated stimulation. A 3-minute resting EEG will be collected from each participant, and they will be instructed not to actively engage in any cognitive or mental activity. In all stimulation sessions, evaluations will be carried out, the evaluated outcomes will be: change in EEG microstates, cognitive function and motor function. Statistical analyzes will be performed using SPSS software (Statistical Package for Social Sciences - SPSS Inc, Chicago IL, USA for Windows, Version 20.0) and MATLAB (9.2.0 (MathWorks, Inc., Natick, MA) with a defined level of significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

- Individuals diagnosed with stroke for more than 6 months;

Proven by means of magnetic resonance imaging or computed tomography;

Individuals aged 18 and over;

Both sexes;

Patients with mild to moderate degree of injury severity (NIHHS < 17 points)

Exclusion Criteria:

- Individuals who are unable to communicate verbally;

Use of drugs that modulate the activity of the Central Nervous System;

Carriers of implanted metallic or electronic devices; cardiac pacemaker;

Habitual use of drugs or alcohol;

Report of history of epilepsy; gestation; people with traumatic brain injury or tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in EEG microstates in each stimulation condition | immediately after the sessions
  Microstate analysis was performed using the EEGLAB microstate plugin developed by Thomas Koenig (Koenig, 2021). First, at the individual level, we compute global field power (GFP) across all channels and microstate segmentation using the modified k-means clustering algorithm method to isolate map topographies. Polarity was ignored during microstate analysis. After obtaining the microstate segmentation of each participant, we calculated an average of the microstate segmentation of each group as models. The successive original individual EEG series were then divided into four classic microstate maps (they are labeled as four classes A, B, C and D, which are left-right direction (type A), left-right direction (type B), anteroposterior direction (type C) and frontocentral maximum (type D)).

SECONDARY OUTCOMES:
Cognitive function - trail test (TMT) A and B | immediately after the sessions
  TMT consists of connecting letters in the order they appear in the alphabet (A tracks); or letters to numbers, also following the sequence in which they appear in the alphabet, for example, 1-A-2-B and so on (B tracks), with the possibility of evaluating the cognitive components of planning, organization, attention, perseverance and memory.
Cognitive function - clock drawing test | immediately after the sessions
  Currently, the RDT is widely used, it is simple to apply and quick to perform, which assesses several cognitive dimensions, such as memory, motor function, executive function and verbal comprehension. Regarding its score, the Shulman scale scores 5 points in total and a cut-off point equal to 3. The Mendez scale scores up to 20 points for the perfect design of the watch, with a cut-off point equal to 18 points.
Cognitive function - verbal fluency test (VF). | immediately after the sessions
  The VF test assesses several domains such as working memory, language, organizational skills and sequencing. In this test, the patient is asked to speak the largest number of words (within each required category). In the VF test, responses are scored, but repetitions are not considered.
motor function | immediately after the sessions
  The Timed Up and Go Test (TUG) test will be used

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Dra, Principal Investigator — Federal University of Paraiba
Locations (1):
- Aging and Neuroscience Studies Laboratory, João Pessoa, Brazil

IPD SHARING:
Plan to Share IPD: No